CLINICAL TRIAL: NCT03666039
Title: Reversing Maladaptive Reorganization in Frail Brains: Sensorimotor Training, Brain Plasticity and the Role of Brain-derived Neurotrophic Factor
Brief Title: Reversing Maladaptive Reorganization in Frail Brains
Acronym: FRAILBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Prof Herta Flor, Scientific Director, Prof. Dr. Dr. h.c., Central Institute of Mental Health, Mannheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FRAILBRAIN
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Neuroplasticity; Sensorimotor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor training (Experimental): The participants will receive a tablet-based app for at home training that contains sensorimotor components.
  Interventions: Behavioral: Trainings app
- Control training (Active Comparator): The participants will receive a tablet-based app for at home training that contains relaxing components.
  Interventions: Behavioral: Trainings app

INTERVENTIONS:
Behavioral: Trainings app — Sensorimotor trainings app for at home Training (tablet-based)

SUMMARY:
Neuroscientific models of maladaptive aging emphasize the loss of sensorimotor stimulation and reduced modulatory capacities as core processes in the development of maladaptive plastic changes of the brain and subsequent cognitive and bodily decline as determinants of frailty and multimorbidity in old age. The investigators plan to analyze anatomical, neurophysiological, and neuropsychological correlates of maladaptive plasticity in frail persons and plan to test how innovative interventions that target maladaptive plasticity alter brain function and neurocognitive skills. There are novel interventions that have been shown to target the neurocognitive deficits and enhance plasticity in brain areas that are affected first in the progress of aging. Specifically, sensory training has been employed to enhance relevant input to the brain and to improve neuromodulatory function and has yielded high effect sizes. The investigators will perform proof of concept studies to examine the utility of sensorimotor training and examine the role of brain-derived neurotrophic growth factor to enhance brain plasticity and memory functions, as well as their transfer to other cognitive domains. The investigators will implement motivational enhancement strategies using virtual reality in these treatments that can further boost training effects and plasticity, but have not been employed in these treatments so far. Biomarkers for the remediation of maladaptive changes will involve neuropsychological assessments, brain imaging, brain-derived neurotrophic factor (BDNF) levels, and BDNF genotype. Thus, the investigators will be able to comprehensively characterize dysfunctional plasticity and the specific mechanisms of the interventions that are employed and investigate innovative clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Frail individuals (Fried criteria)

Exclusion Criteria:

* Alzheimer or strong cognitive/dementia impairments, strong neurological impairments, age below 65

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Neuroplasticity measures of brain Imaging I: brain responses at rest and task-based (sensorimotor) | 2 months
  Blood oxygenation level dependent (BOLD) signal changes
Body parameter: weight and height | 2 months
  Information on weight and height will be combined to report BMI in kg/m^2
Body parameter: muscles | 2 months
  Muscle strength in electromyogram amplitudes
Neuroplasticity measures of brain Imaging: brain size | 2 months
  Volume of different brain regions
Neuroplasticity measures of brain Imaging: brain diffusion | 2 months
  Brain diffusion in fractional anisotropy values

SECONDARY OUTCOMES:
Well-being | 2-3 months
  Questionnaire data on mood and mental health will be standardized and integrated into one mean score of well-being (computation of a mean values across the questionnaire scores)
Cognitive health | 2-3 months
  Behavioral performance data during cognitive testing will be standardized integrated into one mean score of cognitive functioning (computation of a mean value across response times in the cogniitve tests)

CONTACTS AND LOCATIONS:
Locations (1):
- CIMH - Department of Cognitive and Clinical Neuroscience, Mannheim, Germany

REFERENCES:
- [Derived] Beier F, Loffler M, Nees F, Bekrater-Bodmann R, Silvoni S, Desch S, Loffler A, Hausner L, Frolich L, Flor H. Effects of an app-based sensorimotor training in promoting neuroplasticity and neuropsychological functioning in frailty: A randomized controlled trial. Arch Gerontol Geriatr. 2023 Dec;115:105202. doi: 10.1016/j.archger.2023.105202. Epub 2023 Sep 17. PMID 37776754
- [Derived] Beier F, Loffler M, Nees F, Hausner L, Frolich L, Flor H. Sensory and motor correlates of frailty: dissociation between frailty phenotype and frailty index. BMC Geriatr. 2022 Sep 15;22(1):755. doi: 10.1186/s12877-022-03416-6. PMID 36109693
- [Derived] Beier F, Loffler M, Nees F, Hausner L, Frolich L, Flor H. Promoting neuroplasticity and neuropsychological functioning in frailty through an app-based sensorimotor training: study protocol for a randomized trial. BMC Geriatr. 2021 Jun 3;21(1):343. doi: 10.1186/s12877-021-02293-9. PMID 34082710